CLINICAL TRIAL: NCT02258854
Title: An Open-Label, Non-Randomized, Single-Arm, Rollover Study to Continue Dosing of Gevokizumab in Subjects With Non Infectious Intermediate-, Posterior-, or Pan-Uveitis Patients Who Each Successfully Completed Either the X052130/CL3-78989-005 (EYEGUARD™-A) or the X052131/CL3-78989-006 (EYEGUARD™-C) Study or Who Have Controlled Ocular Inflammation After Receiving Study Drug in Study X052133 (EYEGUARD™-US)
Brief Title: An Open-label, Rollover Study Providing Continued Dosing of Gevokizumab in Order to Assess Long-term Gevokizumab Safety Data
Acronym: EYEGUARD™-E
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: XOMA (US) LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X052132
Record Dates: First submitted 2014-10-02; First posted 2014-10-08 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Uveitis
Keywords: Uveitis; Non-infectious Uveitis; Intermediate Uveitis; Posterior Uveitis; Panuveitis; Behçet's disease uveitis
MeSH Terms: conditions — Uveitis; Uveitis, Intermediate; Uveitis, Posterior; Panuveitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose 2 gevokizumab (Experimental)
  Interventions: Drug: Dose 2 gevokizumab

INTERVENTIONS:
Drug: Dose 2 gevokizumab — Solution for subcutaneous injection

SUMMARY:
The purpose of this study is to provide continued dosing of gevokizumab in order to obtain and assess long-term gevokizumab safety data.

ELIGIBILITY:
Inclusion Criteria:

* Completed either the X052130/CL3-78989-005 or the X052131/CL3-78989-006 study's masked D392 or OL-224 completion day visits or had controlled ocular inflammation after having received study drug in Part 2 of study X052133

Exclusion Criteria:

* Discontinued from the previous study

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-03; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent Adverse Events | 108 weeks

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - Chandler, Arizona
  - Phoenix, Arizona
  - Beverly Hills, California
  - Redlands, California
  - Riverside, California
  - Sacramento, California
  - Santa Ana, California
  - Victorville, California
  - Golden, Colorado
  - Littleton, Colorado
  - Bridgeport, Connecticut
  - Lakeland, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Ellsworth, Maine
  - Baltimore, Maryland
  - Cambridge, Massachusetts
  - Waltham, Massachusetts
  - Jackson, Michigan
  - Royal Oak, Michigan
  - Omaha, Nebraska
  - Bloomfield, New Jersey
  - Teaneck, New Jersey
  - Belmont, North Carolina
  - Charlotte, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia